CLINICAL TRIAL: NCT02684708
Title: European Network-Paediatric Hodgkin Lymphoma Study Group (EuroNet-PHL) Second International Inter-Group Study for Classical Hodgkin Lymphoma in Children and Adolescents
Brief Title: Second International Inter-Group Study for Classical Hodgkin Lymphoma in Children and Adolescents
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Giessen (Other)
Collaborators: Deutsche Krebshilfe e.V., Bonn (Germany) (Other); Euronet Worldwide (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EuroNet-PHL-C2
Record Dates: First submitted 2015-11-19; First posted 2016-02-18 (Estimated); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Classical Hodgkin Lymphoma
MeSH Terms: interventions — Cyclophosphamide; Vincristine; Prednisone; Dacarbazine; prednylidene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- COPDAC-28 (Active Comparator): cyclophosphamide, vincristine, prednisone, dacarbazine; cyclophosphamide 500 mg/m2, per infusion on day 1 + 8; vincristine 1.5 mg/m2 intravenously (capping dose 2 mg) on day 1 + 8 and prednisone 40 mg/m2/day by mouth divided into 3 doses (capping dose 80 mg/day) on day 1 - 15 and dacarbazine 250 mg/m2 infusion on day 1 - 3
  Interventions: Drug: cyclophosphamide, vincristine, prednisone, dacarbazine
- DECOPDAC-21 (Experimental): patients with intermediate and advanced stages will be randomized after the induction therapy to receive either COPDAC-28 standard consolidation or the intensified DECOPDAC-21. cyclophosphamide dose augmented to 625 mg/m2 and adminstered per infusion on day 1 and day 2; vincristine dose not changed; prednisone 40 mg/m2/day by mouth on day 1 - 8 (no capping dose prescribed), i.e. dose-reduction; dacarbazine dose not changed; etoposide infusion100 mg/m2/day on day 1 - 3 and doxorubicine 25 mg/m2 per infusion on day 1as additional drugs in comparison to active comparator; cycle is administered as 21 days instead of 28 days-cycle for intensification
  Interventions: Drug: cyclo, vcr, pred, dacarb,etop and doxo

INTERVENTIONS:
Drug: cyclophosphamide, vincristine, prednisone, dacarbazine — 28-day chemotherapy cycle
  Other Names: CYC, VCR, PRED, DTIC
  Arms: COPDAC-28
Drug: cyclo, vcr, pred, dacarb,etop and doxo — 21-day chemotherapy cycle
  Other Names: CYC, VCR, PRED, DTIC, ETO, DOXO
  Arms: DECOPDAC-21

SUMMARY:
The EuroNet-PHL-C2 trial is an international, multicentre, randomised controlled trial with the aims to reduce the indication for radiotherapy in newly diagnosed patients with classical Hodgkin lymphoma without compromising cure rates and to investigate a chemotherapy intensification randomisation in intermediate and advanced classical Hodgkin lymphoma to compensate for reduction in radiotherapy.

DETAILED DESCRIPTION:
EuroNet-PHL-C2 is a comprehensive treatment strategy for all first line classical Hodgkin Lymphoma (cHL) patients under 18 years (under 25 years in UK, Italy and France). The overall strategy is risk stratified (defining chemotherapy) and response adapted (defining radiotherapy) to tailor the amount of treatment to the individual patient and decrease long term complications.

* Radiotherapy indication will be restricted. Patients with a negative PET scan after two cycles of OEPA chemotherapy (Early Response Assessment - ERA) will not receive radiotherapy. The threshold for negative PET scan at ERA shifts from the previously used Deauville 1 and 2 = negative (as in the C1 trial) to Deauville 1, 2 and 3 = negative, thereby increasing the number of negative patients without indication for RT.
* Chemotherapy Randomisation

All intermediate (TL-2) and advanced stage (TL-3) patients will be randomised between respectively 2 or 4 standard COPDAC-28 or intensified DECOPDAC-21 consolidation chemotherapy cycles. To avoid delayed consolidation, randomisation has to be performed before ERA and as soon as the TL-assignment is confirmed by central review. Therefore two randomised sub-studies arise based on the ERA PET response:

Patients with adequate response at ERA do not receive radiotherapy - a randomised controlled chemotherapy comparison to show that intensified DECOPDAC-21 consolidation chemotherapy improves EFS as compared to standard COPDAC-28

Patients with inadequate response at ERA - a randomised controlled chemotherapy-radiotherapy comparison - to show that DECOPDAC-21 combined with radiotherapy restricted to sites that remain FDG-PET positive at the end of all chemotherapy (Late response assessment - LRA) has comparable EFS compared to COPDAC-28 plus standard involved node radiotherapy as in the C1 trial.

* Risk stratification is refined Former treatment groups (TG) of the EuroNet-PHL-C1 trial are reassigned into treatment levels (TL) by shifting early stage patients (former TG-1) with risk factors into TL-2.
* Semi-quantitative 'qPET' Results of semi-quantitative qPET are formally integrated into the response assessment.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed primary diagnosis of classical Hodgkin's lymphoma
* patients under 18 years of age on the date of written informed consent. In specialized Teenage and Young Adult (TYA) units in France, Italy and UK patients up to under 25 years of age can also be enrolled. Lower age limits will be country specific according to national laws or formal insurance requirements that may preclude very young patients.
* written informed consent of the patient and/or the patient's parents or guardian according to national laws
* negative pregnancy test within 2 weeks prior to starting treatment for female patients with childbearing potential

Exclusion Criteria:

* prior chemotherapy or radiotherapy for other malignancies
* pre-treatment of Hodgkin's lymphoma (except for 7-10 days steroid pre-phase of a large mediastinal tumour)
* diagnosis of lymphocyte-predominant Hodgkin's lymphoma
* other (simultaneous) malignancies
* contraindication or known hypersensitivity to study drugs
* severe concomitant diseases (e.g. immune deficiency syndrome)
* known HIV-positivity
* residence outside the participating countries where long term follow-up cannot be guaranteed
* pregnancy and/or lactation
* patients who are sexually active and are unwilling to use adequate contraception during therapy and for one month after last trial treatment
* current or recent (within 30 days prior to date of written informed consent) treatment with another investigational drug or participation in another interventional clinical trial

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2200 (Estimated)
Dates: Start 2015-10-01; Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Event-free survival | 5 years
  Time from treatment start until relapse/progression, secondary malignancy or death

SECONDARY OUTCOMES:
Overall survival | 5 years
  Time from treatment start until death
Progression-free survival | 5 years
  Time from treatment start until relapse/progression or death
CTC (common toxicity criteria) grading during any individual treatment element including assessment of osteonecrosis | 5 years
  Toxicity assessment according to CTCAE v4.0
Time from day of PET imaging until decision on response category at ERA or LRA, respectively | 5 years
  Quality of Imaging (CT,MRI and PET-CT) acquisition,
Time from last day of chemotherapy to first day of radiotherapy in patients with radiotherapy indication | 5 years
  Quality of chemo-and radiotherapy delivery
Time from last dose of prednisone/prednisolone in OEPA to start of the first consolidation cycle | 5 years
  Quality of chemotherapy delivery

CONTACTS AND LOCATIONS:
Overall Officials: Dieter Koerholz, MD, Study Chair — Justus-Liebig University of Giessen
Locations (19):
- Royal Children's Hospital and Monash Medical Centre Royal Children's Hospital, Victoria Park, Australia
- St. Anna Kinderspital, Vienna, Austria
- Paediatric haemato-oncology, University Hospitals of Leuven, Leuven, Belgium
- Dpt. of Pediatric Hematology and Oncology, Faculty Hospital Motol, Prague, Czechia
- Department of Pediatric Hematology/Oncology (5054) The Child and Youth Clinic, University Hospital of Copenhagen, Copenhagen, Denmark
- Service d'Oncohématologie, Hopital d'Ènfants Armand Trousseau, Paris, France
- Justus Liebig University of Giessen, Giessen, Germany
- Our Lady's Children's Hospital, Crumlin, Dublin, Ireland
- Tel Aviv University Schneider Children's Medical Center of Israel The Rina Zaizov Pediatric Hematology Oncology Division, Petah Tikva, Israel
- Pediatric Radiotherapy and Youth Area Unit C.R.O. - Centro di Riferimento Oncologico IRCCS, Aviano, Italy
- Princess Máxima Center for pediatric oncology, Utrecht, Netherlands
- Starship Blood and Cancer Centre, Starship Children's Hospital, Auckland, New Zealand
- Department of Medical Oncology Oslo University Hospital, Oslo, Norway
- Head of Department of Pediatric Oncology and Hematology, Polish-American Pediatric Institute, Jagiellonian University Medical Faculty, Krakow, Poland
- Clinic of Pediatric Oncology University Children's Hospital, Bratislava, Slovakia
- Sección de Onco-Hematología Pediátrica Hospital Universitario Virgen Macarena y Virgen del Rocío, Seville, Spain
- Pediatric Hematology & Oncology Children´s University Hospital, Uppsala, Sweden
- CHUV - Centre Hospitalier Universitaire Vaudois = LS, Départment femme - meré - enfant, Service de pédiatrie, Unité d'hématologie-oncologie pédiatrique, Lausanne, Switzerland
- University College London Hospitals, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pabari R, McCarten K, Flerlage J, Lai H, Mauz-Korholz C, Dieckmann K, Palese M, Kaste S, Castellino SM, Kelly KM, Stoevesandt D, Kurch L. Hodgkin lymphoma involving the extra-axial CNS: an AHOD1331, PHL-C1, and PHL-C2 report from the COG and EuroNet-PHL. Blood Adv. 2024 Sep 24;8(18):4856-4865. doi: 10.1182/bloodadvances.2023012346. PMID 39058968
- [Derived] Drechsel KCE, Pilon MCF, Stoutjesdijk F, Meivis S, Schoonmade LJ, Wallace WHB, van Dulmen-den Broeder E, Beishuizen A, Kaspers GJL, Broer SL, Veening MA. Reproductive ability in survivors of childhood, adolescent, and young adult Hodgkin lymphoma: a review. Hum Reprod Update. 2023 Jul 5;29(4):486-517. doi: 10.1093/humupd/dmad002. PMID 36779325
- See also: Hodgkin lymphoma treatment in children and adolescents — https://www.clinicaltrialsregister.eu/ctr-search/search?query=EuroNet-PHL-C2